CLINICAL TRIAL: NCT05151380
Title: Evaluation Clinique Et Cyto-histologique Du Traitement Laser CO2 Fractionné Sur Les Syndromes Génito-Urinaires De La Ménopause Liés À L'atrophie Vaginale
Brief Title: Clinical and Cyto-histological Evaluation of Fractional CO2 Laser Treatment on Genito-Urinary Syndromes of Menopause Related to Vaginal Atrophy
Acronym: ATROVENANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A01625-36
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Genitourinary Syndrome of Menopause

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Women with CO2 laser MonaLisa Touch ® sessions (Other): Women with 3 sessions of CO2 laser MonaLisa Touch ®
  Interventions: Device: CO2 laser MonaLisa Touch ®

INTERVENTIONS:
Device: CO2 laser MonaLisa Touch ® — 3 sessions of SmartXide fractional CO2 laser via the MonaLisa Touch® device, spaced 4 weeks apart, will be performed. An additional comfort session will be performed at 1 year if needed.
  The handpiece of the MonaLisa Touch® device is applied to the vaginal walls with a 360° scan, between 800 and 1100µs, to the vaginal orifice

SUMMARY:
Estrogen deficiency can occur naturally during menopause or as a secondary effect of various treatments for breast or pelvic cancer and can lead to very disabling vulvovaginal symptoms, since it is associated with an anatomical and functional cellular modification of the urogenital sphere. These changes result in urogenital atrophy responsible for vaginal dryness, painful intercourse (dyspareunia), discomfort, itching and burning sensations, dysuria, urgency and incontinence. These symptoms, which significantly affect quality of life, are found in more than 40% of menopausal women and are grouped under the term Genitourinary Syndrome of Menopause (GSM). General or local estrogen-based treatments improve patients' symptoms, but remain contraindicated in women who have had breast cancer. Non-estrogenic local treatments are less effective, remain restrictive and are therefore often abandoned.

The CO2 laser is currently part of the therapeutic arsenal for the management of patients with GSM. This device prevents and eliminates the effects of low estrogen levels on vaginal tissue by restoring the characteristic conditions of the vaginal mucosa of a woman of childbearing age. This simple treatment, which lasts only a few minutes, is safe and painless and has no serious side effects. It restores the tone and elasticity of the tissues, with positive effects on the quality of life and the couple's relationship. The investigators wish to evaluate the possible changes of the genital sphere in a longitudinal way (before, during and after the treatment), including the induced cytohistological changes, in patients with GSM who can benefit of this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women over 40 years of age
* Patients with natural menopause or menopause secondary to cancer treatment (breast, pelvis or other)
* Patients with vaginal and/or urinary, non-vulvar GSM
* Patients for whom CO2 laser therapy is proposed

Exclusion Criteria:

* Vulvovaginal infections (vaginosis)
* Uninvestigated vaginal hemorrhage
* Herpes
* Pregnancy or breastfeeding
* Cervico-vaginal pathology (cervical and/or vaginal dysplasia)
* Suspected or diagnosed HPV
* Significant vaginal prolapse
* Patients on hormone replacement therapy

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
The main objective of the study is to analyze the evolution of GSM by the use of the MonaLisa Touch ® fractionated laser. | 3 months
  The primary endpoint is the comparison of the patient's clinical score composed of a visual analogic scale measuring the intensity of symptoms related to vaginal atrophy (i.e., vaginal burning, vaginal pruritus, vaginal dryness, dyspareunia, and dysuria), before and after 3 laser sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche-Comté, Trévenans, France

IPD SHARING:
Plan to Share IPD: No